CLINICAL TRIAL: NCT05034731
Title: Evaluation of Remote Fitting in Adult and Pediatric Users of the HiResolution Bionic Ear System
Status: Completed | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR0121
Record Dates: First submitted 2021-07-28; First posted 2021-09-05 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss; Ear Diseases; Hearing Disorders; Otolaryngological Disease
MeSH Terms: conditions — Hearing Loss; Ear Diseases; Hearing Disorders; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Electric Only (Other)
  Interventions: Device: Remote Fitting; Device: In-Office Fitting
- Aidable Residual Hearing (Other)
  Interventions: Device: Remote Fitting; Device: In-Office Fitting

INTERVENTIONS:
Device: Remote Fitting — Processors will be programmed using remote fitting application.
Device: In-Office Fitting — Processors will be programmed using standard Target CI application.

SUMMARY:
This is a prospective within-subjects repeated-measures study that will enroll 17 users 13 years or older implanted with a HiResolution Bionic Ear System.

DETAILED DESCRIPTION:
The overall goal of this clinical study is to demonstrate the safety and efficacy of the remote fitting option. Hearing outcomes are expected to be similar whether a study subject's sound processor is programmed in the traditional method in the audiologist's office or whether programming is performed via remote fitting. Therefore, the study described herein uses a non-inferiority design to determine whether sentence recognition in quiet is no worse with remote fitting than in an in-office setting.

ELIGIBILITY:
Inclusion Criteria All Subjects

* Ability to provide Informed Consent/Assent
* 13 years of age or older
* Unilateral or bilateral user of a HiResolutionTM Bionic Ear System (HiRes 90KTM, HiRes 90KTM Advantage, HiResTM Ultra, HiResTM Ultra 3D)
* Minimum of 6 months of CI experience with a minimum of 1 month experience with a Naída CI or Sky CI sound processor
* At least moderate open-set speech recognition abilities (defined as speech in quiet score ≥ 60% as assessed at Visit 1)
* Minimum average score ≥ 3 on the Mobile Device Proficiency Questionnaire (MDPQ-16)
* English language proficiency as determined by the Investigator
* Willingness to use a BTE sound processor for the duration of the study

Inclusion Criteria Specific to Aidable Residual Hearing Group

* Residual low frequency hearing sensitivity (pure tone average of < 70 dB HL for 125, 250, and 500 Hz) and a severe-to-profound high-frequency sensorineural hearing loss (pure tone average of ≥ 70 dB HL for 1,000, 2,000, 3000, 4,000, and 8,000 Hz) in the implanted ear for unilaterally implanted subjects and in both ears for bilaterally implanted subjects
* Willingness to use an in-canal acoustic earhook for the duration of the study

Exclusion Criteria:

* Clinical presentation indicative of potential implanted device malfunction
* Unrealistic expectations regarding potential benefits, risks and limitations of the investigational device as determined by the Investigator
* Unwillingness or inability of subject to comply with all investigational requirements as determined by the Investigator

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigators recruited study subjects from their clinical practices. The first patient visit occurred on 08/18/21 and last patient visit occurred on 05/23/22. Of the 19 enrolled, 2 were deemed ineligible to continue after visit 1 and 17 subjects were assigned to a study; 12 subjects were enrolled in the EO group and 5 subjects were enrolled in the ARH sub-group based on the results of their audiometric testing. All 17 subjects completed the study, with no withdrawals or losses to follow up.
Pre-assignment Details: Per protocol, a subject is considered enrolled upon giving written informed consent. After undergoing the ICF process, subjects completed a hearing test. Depending on the outcome of that test, eligible subjects were enrolled for aidable residual hearing (ARH) fitting with an acoustic earhook. Unilaterally implanted subjects not meeting ARH fitting criteria were enrolled for electric only (EO) fitting. Bilaterally implanted subjects meeting ARH criteria only in one ear were screen failed.
Groups:
- Electric Only (EO): Any subject that did not meet the ARH fitting criteria was enrolled in the EO fitting group. The EO group were fit with the investigational processor and an Advanced Bionics T-mic for the duration of the study. All subjects (both EO and ARH) underwent the same testing procedures after appropriately fitted.
- Aidable Residual Hearing (ARH): A group of subjects that met the general study criteria and the inclusion criteria for ARH as follows:
  * Residual low frequency hearing sensitivity (pure tone average of < 70 dB HL for 125, 250, and 500 Hz) and a severe-to-profound high-frequency sensorineural hearing loss (pure tone average of ≥ 70 dB HL for 1,000, 2,000, 3000, 4,000, and 8,000 Hz) in the implanted ear for unilaterally implanted subjects and in both ears for bilaterally implanted subjects
  * Willingness to use an in-canal acoustic earhook for the duration of the study
Period: Overall Study
Arm/Group | Electric Only (EO) | Aidable Residual Hearing (ARH)
Started | 13 | 6
Completed | 12 | 5
Not Completed | 1 | 1
Not completed — Screen fail | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Electric Only: Any subject that did not meet the ARH fitting criteria was enrolled in the EO fitting group. The EO group were fit with the investigational processor and an Advanced Bionics T-mic for the duration of the study. All subjects (both EO and ARH) underwent the same testing procedures after appropriately fitted.
- Aidable Residual Hearing (ARH): Includes subjects that met all general inclusion criteria and hearing inclusion criteria specific for ARH group.
  * Residual low frequency hearing sensitivity (pure tone average of < 70 dB HL for 125, 250, and 500 Hz) and a severe-to-profound high-frequency sensorineural hearing loss (pure tone average of ≥ 70 dB HL for 1,000, 2,000, 3000, 4,000, and 8,000 Hz) in the implanted ear for unilaterally implanted subjects and in both ears for bilaterally implanted subjects
  * Willingness to use an in-canal acoustic earhook for the duration of the study
- Total: Total of all reporting groups
Arm/Group | Electric Only | Aidable Residual Hearing (ARH) | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 48.2 [15 to 84] | 66.2 [60 to 78] | 53.8 [15 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 5 | 1 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Speech Performance in Quiet After Chronic Use (EO Only)
Description: The primary efficacy endpoint is the chronic AzBio sentence recognition scores in quiet captured two-to-three weeks post investigational remote fitting (visit 3) as compared to the chronic AzBio sentence recognition scores in quiet captured two-to-three weeks post control in-office fitting (visit 2). Scores are determined on a scale of 0% to 100% words correct with higher scores indicating a better outcome.
Time Frame: 2-3 weeks after fitting
Measure: Mean (Standard Deviation); unit: percentage of correctly recognized words
Arm/Group | Electric Only (EO)
Number analyzed (Participants) | 12
percentage of correctly recognized words
  In-Office Fitting Speech Perception score | 89.28 (3.489)
  Remote Fitting Speech Perception score | 91.94 (2.760)
Statistical Analysis 1: Comparison: Electric Only (EO); Test type: Non-Inferiority — Non-inferiority analyses were based on paired t-tests looking at the differences in speech scores calculated using the investigational speech scores minus the control speech scores. The primary efficacy analyses tested the null hypothesis (inferiority) that the mean of the paired differences in AzBio sentence scores in quite (remote fitting - in-office fitting) are less than or equal to -10 percentile points; p < 0.0001, t-test, 1 sided

2. Primary Outcome: Speech Performance in Quiet - Chronic Use (Includes Overall - Both Groups)
Description: as for outcome 1
Time Frame: Test performed 2-3 weeks after fitting
Measure: Mean (Standard Deviation); unit: percentage of recognized words
Groups:
- EO Group: Any subject that did not meet the ARH fitting criteria was enrolled in the EO fitting group. The EO group were fit with the investigational processor and an Advanced Bionics T-mic for the duration of the study. All subjects (both EO and ARH) underwent the same testing procedures after appropriately fitted.
- ARH Group: Includes subjects that met all general inclusion criteria and hearing inclusion criteria specific for ARH group.
  * Residual low frequency hearing sensitivity (pure tone average of < 70 dB HL for 125, 250, and 500 Hz) and a severe-to-profound high-frequency sensorineural hearing loss (pure tone average of ≥ 70 dB HL for 1,000, 2,000, 3000, 4,000, and 8,000 Hz) in the implanted ear for unilaterally implanted subjects and in both ears for bilaterally implanted subjects
  * Willingness to use an in-canal acoustic earhook for the duration of the study
- Overall (Both Groups): This group includes both the EO and ARH subjects that met inclusion criteria and fitted with an investigational device.
Arm/Group | EO Group | ARH Group | Overall (Both Groups)
Number analyzed (Participants) | 12 | 5 | 17
percentage of recognized words
  In-Office fitting Evaluation | 89.28 (12.088) | 88.46 (8.855) | 89.04 (10.964)
  Remote Fitting Evaluation | 91.94 (9.562) | 88.72 (6.007) | 90.99 (8.613)
Statistical Analysis 1: Comparison: Overall (Both Groups); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: AEs were recorded and tracked between completion of the informed consent form and two weeks after the participant completes the study. This total time period is approximately 6-8 weeks dependent on the subject scheduled visits.
Arm/Group | Electric Only | Aidable Residual Hearing
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5
Other Adverse Events (participants affected / at risk) | 2/12 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electric Only (N=12) | Aidable Residual Hearing (N=5)
Device Implant Failure - Right ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Migraine Headache (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees to submit any publication to Sponsor at least 30 days before submission. Within 30 days, Sponsor advises PI in writing of any information contained therein which is Confidential Information (other than Study Data) or which may impair availability of patent protection for Inventions.

Sponsor has the right to require PI to remove specifically identified CI and/or to delay the publication for an additional 60 days to enable Sponsor to seek patent protection for Inventions.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT05034731/Prot_SAP_000.pdf